CLINICAL TRIAL: NCT00356902
Title: Effect of Titrating Oxygen Concentration During Resuscitation of the Newborn on Achieving Normoxemia
Brief Title: Comparison of Different Oxygen Delivery Strategies During Resuscitation of Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital (Other); Masimo Corp - Equipment loan (Unknown); Datex Ohmeda - Equipment loan (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT732656
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-09

CONDITIONS: Prematurity; Oxidative Injury; Respiratory Distress
MeSH Terms: conditions — Premature Birth; Dyspnea

INTERVENTIONS:
Procedure: titration of oxygen during resuscitation

SUMMARY:
Preterm infants are born with immature lungs and often require help with breathing shortly after birth. This currently involves administering 100% oxygen. Unfortunately, delivery of high oxygen concentrations leads to the production of free radicals that can injure many organ systems. Term and near-term newborns deprived of oxygen during or prior to birth respond as well or better to resuscitation with room air (21% oxygen) compared to 100% oxygen. However, a static concentration of 21% oxygen may be inappropriate for preterm infants with lung disease. Our study will investigate how adjusting the amount of oxygen given to sick preterm newborns will affect the ability to maintain a safe oxygen level in their blood. Each infant will be assigned to receive one of three treatments at birth. Resuscitation will either start with 21% oxygen and be increased if needed, 100% oxygen and be decreased if needed or 100% oxygen with no changes made (current standard of treatment). The first two groups will have adjustments in oxygen concentration as needed to reach a safe target range of blood oxygen saturation. We anticipate that preterm newborn infants resuscitated with higher oxygen concentrations will have higher than "normal" levels of oxygen in their blood while those resuscitated initially with lower concentrations of oxygen will be more likely to have "normal" oxygen levels in their blood. All premature infants will have a surface probe placed on the right hand to measure the saturation of blood with oxygen. Following the resuscitation, treatment will proceed as per standard of care until hospital discharge. All infants will be admitted to the neonatal intensive care unit given their prematurity. The purpose of this study is to investigate how safely restricting the amount of oxygen delivered to newborns during resuscitation will affect the amount of oxygen in their blood.

Hypothesis: In this randomized control trial, infants resuscitated with a "low oxygen delivery (LOD)" strategy (initiation of resuscitation with 21% O2) will remain normoxemic for the greatest proportion of time during resuscitation and infants resuscitated with a "high oxygen delivery (HOD)" strategy (100% O2 used for the entire resuscitation) will be normoxemic for the smallest proportion of time during resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* inborn
* <= 32 weeks gestation
* respiratory support needed during resuscitation. Respiratory support is defined as provision of continuous positive airway pressure or positive pressure ventilation delivered via either a face mask or an endotracheal tube.

Exclusion Criteria:

* lethal anomalies
* cyanotic congenital heart disease
* known hemoglobinopathy
* risk of persistent pulmonary hypertension

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 215 (Estimated)
Dates: Start 2005-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Proportion of time spent in normoxemia (85-92%)during resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Yacov Rabi, MD, FRCPC, Principal Investigator — University of Calgary; Wendy H Yee, MD, FRCPC, Principal Investigator — University of Calgary; Sophie Y Chen, MD, MSc, Principal Investigator — University of Calgary; Nalini Singhal, MD, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada